CLINICAL TRIAL: NCT04964349
Title: Efficacy of Jessener Solution Versus Intralesional Steroid in Treatment of Alopecia Areata
Acronym: AA
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ahmed Rashad Elshahid, professor of dermatology, venereology and andrology, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Alazhar faculty of medicine; Ahmed Kadah (Other: Alazhar faculty of medicine); Eman Abd-ellatif (Other: Alazhar faculty of medicine)
Record Dates: First submitted 2021-07-13; First posted 2021-07-16 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Intervention Model Description: there are 2 patches of alopecia areata in the same patient one treated with intralesional injection of corticosteroid and the other one will be treated by jessenersolution
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intralesional cortisosteroid injection (Experimental): Intralesional corticosteroid injection
  Interventions: Drug: Corticosteroids Acting Locally
- jessener solution (Experimental): topical jessener solution
  Interventions: Drug: Corticosteroids Acting Locally

INTERVENTIONS:
Drug: Corticosteroids Acting Locally — topical application of jessener solution
  Other Names: topical jessener solution

SUMMARY:
Alopecia areata is believed to be an autoimmune disease. Treatment primarily relies on intralesional and topical corticosteroids. This study was conducted to evaluate Jessener Solutionas a potential therapeutic modality of Alopecia Areataversusintralesional steroid as regards the efficacy, safety, tolerability, and patients' satisfaction.

DETAILED DESCRIPTION:
Background Alopecia areata is believed to be an autoimmune disease resulting from a breach in the immune privilege of the hair follicles causing non scarring hair loss.Treatment primarily relies on intralesional and topical corticosteroids.Up till now, there is nouniversally proven therapy that induces and maintains remission of Alopecia Areata in all patients.

Aims The Aim of Study is to evaluate the efficacyof Jessener solution versus intralesional steroid in treatment of Alopecia Areata.

Patients and Methods The study will include 40 patients diagnosed clinically and dermoscopically as Alopecia Areata with more than two patches of alopecia areata were included. Two treatment modalities with intralesional corticosteroid and topical Jessener Solutionas were performed in two randomly selected patches. Three sessions were done, 3 weeks apart and were followed-up for three months. Evaluation was done using Mac Donald Hull and Norris grading system , Serial photographs and dermoscopic , trichoscopic examination every month will be done and patient will be score.

ELIGIBILITY:
Inclusion Criteria:

* 1.Alopecia Areatamultilocuolaris.2.Age from18-50years old. 3.Wash out period is two months. 4.Ophiasis pattern alopecia areata.

Exclusion Criteria:

* Age less than 12 yearsand more than 40years old. 2.Patient under treatment.3.Patients having another dermatological condition affecting thescalpas eczema.4.Patients with psychiatric disorders.5.Pregnant and lactating females.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-04-21 (Actual); Primary Completion 2021-10-21 (Estimated); Study Completion 2021-11-20 (Estimated)

PRIMARY OUTCOMES:
Effecacy of topical jessener solution in treatment of alopecia areata | 6 monthes
  Effecacy of topical jessener solution in treatment of alopecia areata

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elshahid, MD, Study Chair — Alazhar faculty of medicine
Locations (1):
- Alazhar faculty of meidicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No